CLINICAL TRIAL: NCT06569654
Title: Effectiveness of Task-Oriented Rehabilitation With SaeboFlex Splint on Independence, Visual Motor Skills, and Depression in Stroke Patients: A Randomized Controlled Study
Brief Title: Task-Oriented Rehab With SaeboFlex: Impact on Independence, Visual Motor Skills, and Depression in Stroke Patients
Acronym: Randomized
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Başar Öztürk, Assoc. Prof., Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fztbasarozturk
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Depression; Splints
Keywords: Occupational therapy; Activities daily living; Neurorehabilitation
MeSH Terms: conditions — Stroke; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group received additional task-oriented repetitive training using the SaeboFlex orthosis, a dynamic wrist-hand-finger orthosis designed to facilitate upper limb rehabilitation in stroke participants. The SaeboFlex orthosis is a custom-fabricated, non-electric mechanical device that assists participants with significant upper extremity weakness, particularly those without active finger extension, in performing repetitive task practice
  Interventions: Device: Saebo splint
- Control group (No Intervention): Both the control and intervention groups received regular rehabilitation, which included physical therapy, occupational therapy and visual cognitive rehabilitation.
  During the regular rehabilitation program, participants received a comprehensive range of therapies aimed at improving their overall functional abilities and quality of life. The key components of the regular rehabilitation included:

INTERVENTIONS:
Device: Saebo splint — The SaeboFlex orthosis was fitted individually for each participant in the intervention group. The orthosis was adjusted to ensure proper alignment and comfort.
  Participants were instructed on how to don and doff the orthosis correctly and safely.
  The orthosis positions the wrist and fingers in extension in preparation for grasp and release activities, enabling participants to perform functional tasks despite limited voluntary movement.
  Task-Oriented Repetitive Training:
  The intervention consisted of 45-minute sessions, conducted twice a week, over a period of 12 weeks.
  Each session focused on repetitive, task-oriented exercises designed to improve motor function and enhance neuroplasticity.
  Training Activities:
  * Moving the Ball
  * Bringing the Ball to the Mouth
  * Reaching Towards a Target
  * Manipulating the Ball Around a Target
  * Placing the Ball into Tubes
  * Throwing the Ball
  * Catching a Rolling Ball
  Other Names: Task-Oriented Repetitive Training
  Arms: Intervention group

SUMMARY:
Objective: The SaeboFlex orthosis is designed to assist individuals with upper extremity weakness in performing repetitive tasks. This study is planned to evaluate its effectiveness in improving upper extremity functions in stroke patients.

Methods: A randomized controlled study is planned to be conducted with 30 stroke patients, who will be divided into a control group (15 patients) and an intervention group (15 patients). The intervention group will receive task-oriented training with the SaeboFlex splint for 12 weeks, twice a week for 45 minutes, in addition to regular rehabilitation. The control group will continue with standard rehabilitation. Planned outcome measures include the Brunnstrom Stages, Stroke Impact Scale, Fugl-Meyer Assessment, Action Research Arm Test, joint range of motion, and Beck Depression Inventory. Non-parametric tests will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Stroke occurrence at least 6 months prior
* Score of 23 or higher on the Standardized Mini Mental Test
* Brunnstrom stage 2 or 3
* Ability to maintain sitting balance
* Active shoulder and elbow flexion of 15 degrees or more
* Wrist extension with finger extension of 15 degrees or more
* Active finger flexion up to 25% of a full fist position

Exclusion Criteria:

* Presence of another neurological, orthopedic, or psychiatric problem causing activity limitation
* Previous use of the method being studied

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Through study completion, an average of 1.5 year
  The ARAT is a widely used, validated, and reliable measure of upper extremity function. It includes four subscales: grip, grasp, pinch, and gross motor movements. The highest total score is 57, indicating the best performance
Joint Range of Motion | Through study completion, an average of 1.5 year
  Goniometry is used to assess joint range of motion of the trunk, and flexion and extension degrees are recorded.
Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) | Through study completion, an average of 1.5 year
  The LOTCA test is used to evaluate individuals' cognitive abilities before and after intervention. It consists of 22 items grouped into two assessments: pre-treatment and post-treatment. The test assesses orientation, visual-spatial perception, visual-motor organization, thinking skills, and attention. Performance on each subtest and total scores are calculated. In our study, we evaluated only the visual-motor organization and visual-spatial perception parameters
Beck Depression Inventory (BDI) | Through study completion, an average of 1.5 year
  This 21-item scale is used to assess the level of depression. Each question is scored from 0 to 3, resulting in a total score ranging from 0 to 63. Scores between 0-13 indicate no depression, 14-24 indicate moderate depression, and scores above 25 indicate severe depression. The scale has been validated and adapted for the Turkish population
Barthel Index (BI) | Through study completion, an average of 1.5 year
  The Barthel Index, developed by Barthel and Mahoney in 1965, is a reliable and valid instrument used to assess individuals' independence in activities of daily living. In this study, the index was used to determine the level of independence in daily activities. The index scores range from 0 to 100, with scores of 0-20 indicating complete dependence, 21-61 indicating severe dependence, 62-90 indicating moderate dependence, 91-99 indicating mild dependence, and 100 indicating independence
Fugl-Meyer Assessment for Upper Extremity | Through study completion, an average of 1.5 year
  This quantitative impairment index measures sensorimotor recovery following stroke based on Twitchell and Brunnstrom's motor recovery stages. The assessment evaluates motor function, balance, sensation, joint range of motion, and pain across five domains. The total score is 226, and the motor score ranges from 0 to 100. The assessment measures reflex movements of the shoulder, elbow, forearm, wrist, hand, hip, knee, and ankle. The highest score for the upper extremity is 66, and for the lower extremity is 34

SECONDARY OUTCOMES:
Brunnstrom Stages | Before intervention for inclusion stage
  This test evaluates motor development in stroke patients and defines it into 6 stages. The absence of voluntary movement is categorized as stage 1 (flaccid stage), while the presence of isolated movements is considered stage 6. Evaluation is performed separately for the upper extremity, lower extremity, and hand
Mini-Mental State Examination (MMSE) | Before intervention for inclusion stage
  This screening test is used to assess the cognitive status of the participants. It consists of 11 items grouped into 5 main categories: orientation, registration, attention and calculation, recall, and language. Scores range from 0 to 30, with higher scores indicating better cognitive function. The validity and reliability of the test have been established in the Turkish population
Stroke Impact Scale (SIS) | Before intervention for inclusion stage
  This scale assesses the perception of post-stroke quality of life by patients or their caregivers. It consists of 8 subscales and 59 questions. Each question is rated on a 5-point Likert scale, indicating the level of difficulty experienced in the past week. Scores range from 0 to 100 for each subscale, and the SIS also includes an evaluation of post-stroke recovery perception using a visual analog scale (0: No recovery, 100: Complete recovery). The scale has been validated and adapted for the Turkish population

CONTACTS AND LOCATIONS:
Locations (1):
- Fenerbahçe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided